CLINICAL TRIAL: NCT02444117
Title: Autism Spectrum Disorders: Clinical and Neurophysiological Evolutions Through a Functional Rehabilitation of Social Communication
Brief Title: Clinical and Neurophysiological Evolutions Through a Functional Rehabilitation of Social Communication in ASD
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-A012740-45
Record Dates: First submitted 2015-02-18; First posted 2015-05-14 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Autistic Disorder
Keywords: neurophysiology
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: functional rehabilitation of social communication

SUMMARY:
This study aims to identify clinical and biological markers which would allow to evaluate precisely the evolution of children with autism spectrum disorders throughout intervention.

DETAILED DESCRIPTION:
200 children with autism spectrum disorders (1-12 years old) will be included in a 2 years follow-up study. Both clinical and neurophysiological evaluations (electrophysiological and eye tracking) will be completed at different times of the follow-up. This integrative approach, combining clinical and biological markers, will allow the identification of different developmental trajectories and then a better individuation of treatment in autism spectrum disorders.

ELIGIBILITY:
Inclusion Criteria:

* re-education of social communication

Exclusion Criteria:

* multi-handicapped associated to ASD

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with autism spectrum disorders
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Clinical changes between Baseline and Two years | 2 years
  Autism Diagnostic Observation Schedule (ADOS)

SECONDARY OUTCOMES:
neurophysiological evaluations at baseline | baseline
  Event related potentials (ERPs) Visual ERPs : P100 evoked by pattern reversing checkerboard stimuli , N170 evoked by faces auditive ERPs: N1c and MMN evoked with an oddball pardaigm using simple tones, MMN evoked with an oddball pardaigm using emotional voices
neurophysiological evaluations at 1 year | 1 year
  Event related potentials (ERPs) Visual ERPs : P100 evoked by pattern reversing checkerboard stimuli , N170 evoked by faces auditive ERPs: N1c and MMN evoked with an oddball pardaigm using simple tones, MMN evoked with an oddball pardaigm using emotional voices
neurophysiological évaluations at 2 years | 2 years
  Event related potentials (ERPs) Visual ERPs : P100 evoked by pattern reversing checkerboard stimuli , N170 evoked by faces auditive ERPs: N1c and MMN evoked with an oddball pardaigm using simple tones, MMN evoked with an oddball pardaigm using emotional voices
Social and cognitive evaluations at baseline | baseline
  Social and Cognitive Evaluation Battery (SCEB),
Social and cognitive évaluations at 1 year | 1 year
  Social and Cognitive Evaluation Battery (SCEB),
Social and cognitive évaluations at 2 years | 1 year
  Social and Cognitive Evaluation Battery (SCEB),
Repetitive behaviors évaluations at baseline | baseline
  Repetitive and Restrictive Behavior Scale (RRBS)
Repetitive behaviors évaluations at one year | 1 year
  Repetitive and Restrictive Behavior Scale (RRBS)
Repetitive behaviors at two years | 2 years
  Repetitive and Restrictive Behavior Scale (RRBS)

CONTACTS AND LOCATIONS:
Overall Officials: Joelle Malvy, MD, PhD, Principal Investigator — University Hospital, Tours
Locations (1):
- University hospital Tours, Tours, France

REFERENCES:
- [Derived] Khanna RK, Kovarski K, Arsene S, Siwiaszczyk M, Pisella PJ, Bonnet-Brilhault F, Batty M, Malvy J. Ophthalmological findings in children with autism spectrum disorder. Graefes Arch Clin Exp Ophthalmol. 2020 Apr;258(4):909-916. doi: 10.1007/s00417-019-04594-7. Epub 2020 Jan 9. PMID 31919663